CLINICAL TRIAL: NCT02082119
Title: Hypofractionated IMRT (VMAT-RA) With Temozolomide for Patients With Newly Diagnosed High Grade Glioma (HGG)
Brief Title: Hypofractionated IMRT With Temozolomide for HGG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Istituto Clinico Humanitas, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1138
Record Dates: First submitted 2013-12-13; First posted 2014-03-10 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Grade Glioma (Experimental): To evaluate safety and feasibility of hypofractionated IMRT in addition to chemotherapy, concomitant and adjuvant, in patients with newly diagnosed High Grade Glioma after biopsy.total dose of 60 Gy/ 4 Gy fraction/15 fractions (BED10 84 Gy) will prescribed to the PTV1; a total dose of 42 Gy/2.8 Gy fraction/15 fractions (BED10 53.76 Gy) will prescribed to PTV2 with SIB.
  Interventions: Radiation: Hypofractionated IMRT

INTERVENTIONS:
Radiation: Hypofractionated IMRT — Hypofractionated IMRT

SUMMARY:
To evaluate safety and feasibility of hypofractionated IMRT in addition to chemotherapy, concomitant and adjuvant, in patients with newly diagnosed HGGs after surgery.

Primary endpoint: progression free survival (PFS), Overall Survival (OS) and Toxicity.

Secondary endpoint: to evaluate Quality of life (QoL) of patients after surgery, concomitant chemoradiotherapy and adjuvant chemotherapy through neuropsychological examination.

DETAILED DESCRIPTION:
We designed a study of a hypofractionated intensity modulated radiation therapy (IMRT), using VMAT RapidArc approach. The potential advantage of this approach is to deliver a more selective irradiation to tumor's target with reducing dose to normal brain and to allow to deliver a higher dose, optimizing the therapeutic window

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Karnosky performance status (KPS) ≥60
* Patients aged >70 years with KPS ≥80
* Histopathologically confirmed of HGG
* Estimated survival ≥ 3 months.
* Multifocal tumor
* Normal liver, Kidney and bone marrow function
* Written informed consent

Exclusion Criteria:

* Prior radiation therapy
* KPS ≤ 60
* Age > 70 years and KPS < 70
* Other primary cancer
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piera Navarria, MD, Study Director — Humanitas Cancer Center
Locations (1):
- Istituto Clinico Humanitas, Milan, Italy

REFERENCES:
- [Background] Reddy K, Damek D, Gaspar LE, Ney D, Waziri A, Lillehei K, Stuhr K, Kavanagh BD, Chen C. Phase II trial of hypofractionated IMRT with temozolomide for patients with newly diagnosed glioblastoma multiforme. Int J Radiat Oncol Biol Phys. 2012 Nov 1;84(3):655-60. doi: 10.1016/j.ijrobp.2012.01.035. Epub 2012 Apr 5. PMID 22483738

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Considering a time of enrollment of 2 years and a follow-up time of 2 years, 82 patients are evaluated from June 2013 to May 2015. Patients with newly diagnosed HGGs underwent hypofractionated IMRT in addition to chemotherapy, concomitant and adjuvant, after biopsy, subtotal or gross total surgical resection.
Period: Overall Study
Arm/Group | High Grade Glioma
Started | 82
Completed | 82
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High Grade Glioma
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants] — Age 18 to 70 years
  Participants
    <=18 years | 0
    Between 18 and 65 years | 60
    >=65 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 52
Region of Enrollment [Number; unit: participants]
  Italy | 82

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined by any of the following: ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids; a significant increase in T2/FLAIR non-enhancing lesions on stable or increasing dose of corticosteroids compared with baseline scan or best response after initial of therapy, not due to comorbid events; the appearance of any new lesions; clear progression of non-measurable lesions; or definite clinical deterioration not attributable to another causes apart from the tumor, or to decrease in corticosteroid dose.
Time Frame: 1 year
Population: Patients with newly diagnosed high grade glioma were analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | High Grade Glioma
Number analyzed (Participants) | 82
Participants | 82
Statistical Analysis 1: Comparison: High Grade Glioma; Test type: Other; p < 0.05, t-test, 1 sided

2. Secondary Outcome: Quality of Life (QoL) of Patients After Surgery, Concomitant Chemo-radiotherapy and Adjuvant Chemotherapy
Description: Quality of life (QoL) of patients after surgery, concomitant chemoradiotherapy and adjuvant chemotherapy is evaluated through neuropsychological examination using the Milano-Bicocca Battery (MIBIB). This battery investigated language, memory, apraxia, including visuo-constructional abilities, executive functions and spatial cognition.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | High Grade Glioma
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes